CLINICAL TRIAL: NCT01517659
Title: Non-Invasive Reduction of Fat in the Inner Thighs With the Zeltiq Coolsculpting System
Brief Title: Non-Invasive Reduction of Fat in the Inner Thighs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZA12-002
Record Dates: First submitted 2012-01-17; First posted 2012-01-25 (Estimated); Results first posted 2020-11-17 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2020-08

CONDITIONS: Body Fat Disorder
Keywords: Cryolipolysis; Fat Reduction

STUDY DESIGN:
Masking Description: Panel of blinded physicians evaluated photos of pre-treatment and post-treatment images. Reviewers were blinded to the time point images were collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Fat Reduction (Experimental): The Zeltiq CoolSculpting System will be used to treat subcutaneous fat on each inner thigh.
  Interventions: Device: The Zeltiq CoolSculpting System

INTERVENTIONS:
Device: The Zeltiq CoolSculpting System — Non-invasive cooling is applied to the treatment area with a defined cooling rate and duration.
  Other Names: Cryolipolysis

SUMMARY:
Evaluate the safety and efficacy of non-invasive fat reduction in the inner thighs with the ZELTIQ CoolSculpting System.

DETAILED DESCRIPTION:
The Zeltiq CoolSculpting System, which reduces subcutaneous fat in specific areas of the body, will be studied for safety and efficacy when used in the inner thigh.

ELIGIBILITY:
Inclusion Criteria

1. Male or female subjects > 18 years of age and < 65 years of age.
2. Subject has clearly visible fat on the inner thighs and in the investigator's opinion, may benefit from the treatment.
3. Subject has not had weight change exceeding 10 pounds in the preceding month.
4. Subject with body mass index (BMI) up to 30. [BMI is defined as weight in pounds multiplied by 703 divided by the square of the height in inches.]
5. Subject agrees to maintain his/her weight (i.e., within 5 pounds) by not making any major changes in his/her diet or lifestyle during the course of the study.
6. Subject has read and signed a written informed consent form.

Exclusion Criteria

1. Subject has had a surgical procedure(s) in the area of intended treatment.
2. Subject has had an invasive fat reduction procedure (e.g., liposuction, abdominoplasty, mesotherapy) in the area of intended treatment.
3. Subject has had a non-invasive fat reduction and/or body contouring procedure in the area of intended treatment within the past 6 months.
4. Subject needs to administer, or has a known history of, subcutaneous injections (e.g., heparin, insulin) into the area of intended treatment within the past month.
5. Subject has a known history of cryoglobulinemia, cold urticaria, or paroxysmal cold hemoglobinuria.
6. Subject has a known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
7. Subject has a history of a bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
8. Subject is taking or has taken diet pills or supplements within the past month.
9. Subject has any dermatological conditions, such as moderate to excessive skin laxity, or scars in the location of the treatment sites that may interfere with the treatment or evaluation (stretch marks is not an exclusion).
10. Subject has an active implanted device such as a pacemaker, defibrillator, or drug delivery system
11. Subject is pregnant or intends to become pregnant in the next 8 months.
12. Subject is lactating or has been lactating in the past 6 months.
13. Subject is unable or unwilling to comply with the study requirements.
14. Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
15. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data, or would pose an unacceptable risk to the subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2014-02-12 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Kilmer, MD, Principal Investigator — Laser and Skin Surgery Center of Northern California
Locations (3):
- United States (3):
  - Laser & Skin Surgery Center of Northern California, Sacramento, California
  - Zel Skin and Laser Specialists, Edina, Minnesota
  - Dallas Plastic Surgery Institute, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zelickson BD, Burns AJ, Kilmer SL. Cryolipolysis for safe and effective inner thigh fat reduction. Lasers Surg Med. 2015 Feb;47(2):120-7. doi: 10.1002/lsm.22320. Epub 2015 Jan 13. PMID 25586980

RESULTS

PARTICIPANT FLOW:
Groups:
- Fat Reduction in Inner Thighs: The Zeltiq CoolSculpting System: Non-invasive cooling is applied to the treatment area with a defined cooling rate and duration.
Period: Overall Study
Arm/Group | Fat Reduction in Inner Thighs
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The population includes eligible participants treated with CoolSculpting in the inner thighs.
Arm/Group | Fat Reduction in Inner Thighs
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 48.1 [35 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Caucasian | 41
  Hispanic | 2
  Others | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Pre-Treatment Images Correctly Identified by Reviewers
Description: Change in the treated vs. untreated areas will be assessed by observation of changes in surface contour and/or fat volume by an independent photo review of pre-treatment and post-treatment images of the treated areas. Reviewers will be practicing dermatologists or plastic surgeons. All reviewers will be blinded to post-treatment vs. baseline untreated area. The order in which images will be presented will be randomized; for each subject placement of the baseline, pre-treatment image will be randomized for each pair of subject images. Reviewers will be asked to select the baseline photos for each subject photo series and record selections on a data collection form. The expected success rate is at least 80% correct identification of pre-treatment images and the majority of physician reviewers (2 out 3) correctly identify 75% of the pre-treatment images.
Time Frame: 16 weeks post-treatment
Population: The per protocol population included all subjects who completed follow-up visits and maintained weight within protocol-defined criteria. Pairs of subject photos (pre-treatment + post-treatment) were presented to blinded reviewers. Reviewers were blinded to time points of photos and the order of photo presentations was randomized.
Measure: Number (95% Confidence Interval); unit: percentage of correct identifications
Units Other Than Participants: photo pairs
Arm/Group | Fat Reduction in Inner Thighs
Number analyzed (Participants) | 42
Number analyzed (photo pairs) | 42
percentage of correct identifications | 90.5 [84.4 to 94.7]

2. Primary Outcome: Safety of the CoolSculpting Device and/or Procedure
Description: The number of device- or procedure related adverse events will be tabulated. Adverse event data are collected continuously throughout the study period from the time of enrollment through the 16 week follow-up visit. At the time of an AE report, each study investigator determines the relationship to the investigational device or the study procedure.
Time Frame: Enrollment through 16 weeks post-treatment
Population: All subjects treated with CoolSculpting were included in the analysis group.
Measure: Number; unit: device-or procedure-related AEs
Arm/Group | Fat Reduction in Inner Thighs
Number analyzed (Participants) | 45
device-or procedure-related AEs | 14

3. Secondary Outcome: Subject Satisfaction
Description: Subject satisfaction as assessed by questionnaires administered at 16 weeks post-treatment.
Time Frame: 16 weeks post-treatment
Population: The analysis population included all subject responses collected at the 16 week follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Fat Reduction in Inner Thighs
Number analyzed (Participants) | 45
Participants
  Very to somewhat satisfied w/ procedure and result | 42
  Very visible to somewhat visible fat reduction | 38
  Positive overall effect | 36
  Very likely to somewhat likely to have another tx | 41
  Would recommend CoolSculpting to friend | 40

4. Secondary Outcome: Reduction in Fat Layer Thickness in the Treated Area as Measured by Ultrasound
Description: Change in the fat layer thickness will be calculated by comparison of pre-treatment and 16 week post-treatment ultrasound measurements taken in the area treated with the device, and in the untreated lateral thigh control area. The Sponsor's standardized techniques for obtaining ultrasound imaging will be used. Overall fat layer thickness changes will be normalized for each subject by subtracting the change in the control area from the change in treated area to remove the influence of weight variations. This result is considered the treatment effect. Success is defined as, on average, at least a 1mm or greater reduction in fat layer thickness for the treated region as compared to the untreated control region. Results indicate the fat layer reduction in millimeters.
Time Frame: 16 week-post-treatment
Population: Population includes all subjects with completed ultrasound images and who maintained weight within the protocol-defined weight requirement.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: treated and control sites
Groups:
- Inner Thigh Treated With CoolSculpting: The Zeltiq CoolSculpting System: Non-invasive cooling is applied to the treatment area with a defined cooling rate and duration.
Arm/Group | Inner Thigh Treated With CoolSculpting
Number analyzed (Participants) | 38
Number analyzed (treated and control sites) | 76
mm | -2.8 (2.29)
Statistical Analysis 1: Comparison: Inner Thigh Treated With CoolSculpting; Test type: Other; Mean Difference (Final Values) = 2.61, 95% CI 2-sided [2.23 to 3.27], Standard Deviation 2.29

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from enrollment through the 16 week follow-up visit.
Description: An adverse event is defined as any untoward medical occurrence in a subject, regardless of whether the event is related to the device.
Arm/Group | Fat Reduction in Inner Thighs
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 2/45
Other Adverse Events (participants affected / at risk) | 12/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fat Reduction in Inner Thighs (N=45)
Adrenal gland mass (Endocrine disorders) | 1 (1) — Mass documented 49 days post-treatment. Subsequent laparoscopic adrenalectomy performed. Not related to CoolSculpting procedure or device.
Herniated spinal disc (Musculoskeletal and connective tissue disorders) | 1 (1) — Subject diagnosed with herniated disc 19 days post-treatment. Chronic/long term condition. Not related to CoolSculpting procedure or device.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fat Reduction in Inner Thighs (N=45)
Numbness, persistent numbness (Skin and subcutaneous tissue disorders) | 12 (12) — Mild numbness reported in treatment area. All mild numbness events resolved without medical intervention.
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) — Mild hyper pigmentation at treatment site. Resolution occurred without medical intervention.
Left shoulder injury; capsular tear (Musculoskeletal and connective tissue disorders) | 1 (1) — Shoulder injury sustained during treatment period. Not related to CoolSculpting procedure or device.
Discoloration on soles of feet (Skin and subcutaneous tissue disorders) | 1 (1) — Black pigmented spots reported on soles of feet. Subject had fever with virus prior to report. Resolved 26 days later. Not related to CoolSculpting procedure or device.
Influenza (Infections and infestations) | 1 (1) — Influenza reported during study period. Received 7 day course of antibiotics and symptoms resolved. Not related to CoolSculpting procedure or device.
Seizure (Nervous system disorders) | 1 (1) — Left temporal lobe seizure reported 31 days post-treatment. Determined to be chronic/long term condition. Not related to CoolSculpting procedure or device.
Indentation (Skin and subcutaneous tissue disorders) | 1 (1) — Mild indentation in treated area noted at 16-week follow-up visit. Resolved 29 days after 16-week visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No